CLINICAL TRIAL: NCT02637375
Title: A Pilot Preoperative Trial of Ganetespib With Paclitaxel for Triple-Negative Breast Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never opened (terminated as study drug no longer available)
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB15-0848
Record Dates: First submitted 2015-12-17; First posted 2015-12-22 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: Breast Cancer
Keywords: triple-negative breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — STA 9090; Paclitaxel; Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Therapy (Experimental): Patients will receive ganetespib monotherapy for two weeks followed by twelve weeks of ganetespib/paclitaxel therapy followed by 4 bi-weekly doses of doxorubicin/cyclophosphamide therapy followed by surgery.
  Interventions: Drug: Ganetespib; Drug: Paclitaxel; Drug: Doxorubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Ganetespib
Drug: Paclitaxel
Drug: Doxorubicin
Drug: Cyclophosphamide

SUMMARY:
Based on preclinical data implicating GR, AR, and JAK/STAT activation as potent mechanisms of breast cancer cell survival despite chemotherapy administration (i.e. chemotherapy resistance), the study will test a novel approach for improving chemotherapy effectiveness by adding Hsp90 inhibition to antagonize the anti-apoptotic signaling pathways that are initiated via GR, AR, and JAK/STAT activation.

DETAILED DESCRIPTION:
STUDY OBJECTIVES

Primary:

• To determine tumor GR, AR, JAK and other Hsp90 client protein expression before and after two weeks of ganetespib monotherapy

Secondary:

* To determine the pathological Complete Response (pCR) rate associated with weekly treatment of ganetespib plus paclitaxel followed by the combination treatment of doxorubicin plus cyclophosphamide
* To characterize the toxicity of study treatment

ELIGIBILITY:
Inclusion Criteria:

* Invasive carcinoma of the breast
* ER negative and PR negative tumors defined as < 1% of tumor nuclei that are immunoreactive for ER and PR
* HER2 non-overexpressing status documented as:
* FISH ratio of less than 2.0, OR
* IHC staining of 0 or 1+
* No evidence of distant metastatic disease. Patients with regional lymph node involvement are eligible.
* >18 years old
* Female
* No prior treatment for the disease under study
* No prior treatment within 5 years for any other cancer including chemotherapy, surgery (except for diagnostic biopsy), radiotherapy, hormonal therapy, or investigational agents, unless curative treatment of non-melanoma skin-cancer or in-situ cancer
* Able to understand and sign an informed consent (or have a legal representative who is able to do so)
* Clinically or radiologically measureable disease in the breast after diagnostic biopsy, defined as longest diameter greater than or equal to 2cm
* Willing to undergo three mandatory core biopsies after diagnosis to obtain tissue for biologic expression profiling.
* An Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1
* Adequate bone marrow reserves as evidenced by:
* Leukocytes > 3,000/μL
* Absolute neutrophil count (ANC) > 1,500/μL without the use of hematopoietic growth factors,
* Platelet count > 100,000/μL, and
* Hemoglobin > 9 g/dL
* Adequate hepatic function as evidenced by:
* Serum total bilirubin within institutional normal limits
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase less than or equal to 2.5 × ULN
* Adequate renal function as evidenced by a serum creatinine within ULN or creatinine clearance > 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Eligible for treatment with paclitaxel, doxorubicin and cyclophosphamide
* If of childbearing potential, are willing to abstain from sexual intercourse or to use an effective form of contraception (e.g., a double-barrier method) during the study and for 90 days following the last dose of ganetespib

Exclusion Criteria:

* • Patients may not be receiving any other investigational agents.

  * Patients may not have a known hypersensitivity to any of the components of ganetespib
  * Patients may not have a history of severe allergic reactions to paclitaxel or other drugs formulated in Cremaphor® EL.
  * Patients with a QTc > 470 ms, a family history of long QT Syndrome, and those on medications known to cause Torsades de Pointes will be excluded from the study.
  * Patients may not have an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
  * Patients may not have New York Heart Association (NYHA) Class III or IV congestive heart failure or left ventricular ejection fraction (LVEF) < 50%.
  * As patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study.
  * Patients may not have a need for chronic systemic steroid therapy
  * Patients may not be pregnant or breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in GR protein | 2 weeks

SECONDARY OUTCOMES:
Pathological Complete Response (pCR) rate | 6 month
  Defined as absence of invasive carcinoma in both the breast and axilla at the time of surgery
Ganetespib toxicity | 14 weeks
  Side effects related to Ganetespib as graded per Common Terminology Criteria for Adverse Events (CTCAE) version 4

CONTACTS AND LOCATIONS:
Overall Officials: Rita Nanda, MD, Principal Investigator — University of Chicago